CLINICAL TRIAL: NCT00293943
Title: A Randomized Trial to Investigate the Significance of Complete Versus Incomplete Electrical Isolation of Pulmonary Veins by Radiofrequency-induced Linear Lesions
Brief Title: Randomized Trial of Two Different Strategies to Treat Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: C. R. Bard (Industry); Biosense Webster, Inc. (Industry); Abbott Medical Devices (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFNET-B04-1
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Pulmonary vein ablation; Linear lesions
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Procedure: Pulmonary vein ablation

SUMMARY:
The purpose of this study is to investigate the significance of complete versus incomplete electrical isolation of pulmonary veins by radiofrequency-induced linear lesions in patients with paroxysmal atrial fibrillation.

The study hypothesis ist that the complete linear PV isolation ablation is superior to the non-complete linear PV isolation on the outcome of patients with idiopathic drug-refractory atrial fibrillation. As a second hypothesis in this adaptive study design, the non-inferiority of the complete linear PV isolation strategy will be tested.

DETAILED DESCRIPTION:
Atrial fibrillation can be cured by elimination of triggering events such as atrial extrasystoles originating from the pulmonary veins (PV) by selective or linear radiofrequency current applications.

Although electrical isolation can be demonstrated by a circumferential mapping catheter positioned at the PV ostium, longterm effect of such EP-guided PV isolation procedures achieve about 60-70% of stable sinus rhythm during follow-up even in experienced centers. Re-investigation of symptomatic patients after initially electrically isolated PVs demonstrated a substantial amount of PV reconduction which might explain the arrhythmia recurrence.

Although it was demonstrated that linear lesions for PV isolation is superior to the selective ablation approach, conflicting data exists on the necessity to achieve complete linear lesions. The groups of Pappone et al and Oral et al both published a success rate of more than 90% of patients in sinusrhythm irrespective of the line completeness, which both groups estimated to be reached in only 30% of cases.

Several advantages and disadvantages could advocate for either the complete versus the incomplete ablation strategy: Performing the complete EP-guided linear PV isolation strategy might take longer (mean duration 4.5 hours vs about 2 hours) and could thereby potentially result in a higher risk of procedure-associated complications (air embolism, thrombus formation, perforation). In addition, three transseptal sheaths might increase the risk of tamponade and might aggravate the ability to safely navigate catheters in the left atrium. Certainly, the procedure costs are higher, since in addition to the 3D mapping system two circular mapping catheters are mandatory to facilitate the lesion deployment and avoidance of intra-PV ablation.

In addition, an ablation strategy that does not depend on complete line deployment may be sufficient to achieve stable sinus rhythm. Although, additional linear lesions between the PV isolation segments and towards the mitral annulus as proposed by several centers with incomplete linear PV isolation approaches might not be necessary to achieve stable sinus rhythm. Potential complications such as atrio-esophageal fistula formation could be avoided if no additional lesions eg. along the LA roof would be necessary. Both the costs of the additional material (transseptal sheaths, circular mapping catheters) and the shorter procedure duration (about 2 hours) would be reduced. On the other hand, these costs would be balanced by the reduced number of re-ablation, if incomplete PV isolation would indeed lead to a higher AF recurrence rate.

Since no data exist on the time course of the deployed ablation lines. Do patients with recurrences of AF always have PV reconduction ? Vice versa, it also remains unclear if all patients with stable sinus rhythm do experience this effect based on longterm PV isolation. To assess the significance of the time course of PV isolation, the proposed study protocol consists therefore of an invasive re-evaluation of all primarily ablated pts scheduled after 3 months of follow-up regardless of arrhythmia recurrence to investigate PV conduction properties.

Finally, patients with symptomatic AF who underwent intensified ECG monitoring indicate that the standard clinical procedures (assessment of symptoms and surface ECG recordings at long intervals) are not sufficient to detect recurrent AF. Therefore, daily ECG monitoring is planned in this trial to detect asymptomatic episodes of AF.

The proposed study protocol aims to investigate in prospective, randomized fashion the significance of complete versus incomplete PV isolation by RFC-induced linear lesions. The ablation will be randomized to a linear encircling around the ipsilateral PVs with the endpoint of complete PV isolation proven by two circumferential mapping catheters versus the same ablation procedure which will be terminated instantaneously when total PV isolation occurs, thereby allowing at least one conduction gap along the isolation line. An invasive re-evaluation is scheduled after 3 months for all pts to assess longterm PV conduction properties.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic paroxysmal symptomatic atrial fibrillation refractory to antiarrhythmic therapy
* Age 50 - 85 years
* Patient willing to participate in randomized trial and an invasive follow-up at month 3 (-6)
* Structural normal heart
* Patient willing and able to participate in 12 months follow-up period
* ECG documentation of atrial fibrillation (ECG, Holter, event recorders, etc) for at least one AF event in the prior year (related to symptomatic or asymptomatic episodes) with an average number of one episode per month
* Written informed consent of the patient

Exclusion Criteria:

* Patients who have had previous pulmonary vein ablation procedures Patients with atrial fibrillation secondary to a reversible cause
* Known presence of intracardiac or other thrombi
* Evidence of obstructive lung disease requiring bronchodilator therapy
* Pregnant females or those of child bearing potential who have not had a negative pregnancy test within 48 hours before treatment.
* Other medical illness (i.e. cancer, congestive heart failure) that may cause the patient to be non-compliant with the protocol, confound the data interpretation or is associated with limited life-expectancy (i.e., less than one year)
* History of bleeding diathesis or suspected pro-coagulant state contraindication to anticoagulation therapy
* Hyperthyroidism or hypothyroidism manifested clinically and in laboratory tests (TSH, T3, T4)
* Participation in a clinical trial within the last 30 days. Simultaneous participation in a registry (e.g. project AB1 of the AFNET) is permitted.
* Drug addiction or chronic alcohol abuse
* Legal incapacity, or other circumstances which would prevent the patient from understanding the aim, nature or extent of the clinical trial
* Evidence of an uncooperative attitude

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2006-02; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
- Time to first recurrence of symptomatic AF with duration of more than 30 sec on trans-telephonic ECG monitoring or detection of asymptomatic AF defined as 2 consecutive recordings of AF during a minimum of 72 hours
  Time to first recurrence of symptomatic AF with duration of more than 30 sec on trans-telephonic ECG monitoring or detection of asymptomatic AF defined as 2 consecutive recordings of AF during a minimum of 72 hours

SECONDARY OUTCOMES:
- Time to first occurrence of any documented relapse of atrial fibrillation
  - Time to first occurrence of any documented relapse of atrial fibrillation
- Number and total duration of documented AF episodes
  - Number and total duration of documented AF episodes
- Number of hospitalizations due to atrial fibrillation
  - Number of hospitalizations due to atrial fibrillation
- Number of visits without hospitalization
  - Number of visits without hospitalization
- Number of "serious adverse events of special interest"
  - Number of "serious adverse events of special interest"
- Procedure parameters (duration, fluoroscopy, number of radiofrequency applications)
  - Procedure parameters (duration, fluoroscopy, number of radiofrequency applications)
- Procedural costs (including the costs of re-ablation if AF recurrence occurs)
  - Procedural costs (including the costs of re-ablation if AF recurrence occurs)
- Quality of life
  - Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Günter Breithardt, MD, Principal Investigator — Universität Münster; Karl-Heinz Kuck, MD, Principal Investigator — General Hospital St. Georg, Hamburg; Stephan Willems, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (3):
- Germany (3):
  - General Hospital St. Georg, Department of Cardiology, Hamburg
  - University Cardiac Center, Hamburg
  - University Hospital, Department of Cardiology, Münster

REFERENCES:
- [Derived] Kuck KH, Hoffmann BA, Ernst S, Wegscheider K, Treszl A, Metzner A, Eckardt L, Lewalter T, Breithardt G, Willems S; Gap-AF-AFNET 1 Investigators*. Impact of Complete Versus Incomplete Circumferential Lines Around the Pulmonary Veins During Catheter Ablation of Paroxysmal Atrial Fibrillation: Results From the Gap-Atrial Fibrillation-German Atrial Fibrillation Competence Network 1 Trial. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003337. doi: 10.1161/CIRCEP.115.003337. PMID 26763226
- See also: Homepage of the German Atrial Fibrillation Network — http://www.kompetenznetz-vorhofflimmern.de